CLINICAL TRIAL: NCT01908010
Title: A Multiple-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ABT-354 in Subjects With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Brief Title: Safety, Tolerability, and Pharmacokinetics of ABT-354 in Subjects With Mild-to-Moderate Alzheimer's Disease on Stable Doses of Acetylcholinesterase Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: M13-080
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1, low dose (Experimental): ABT-354
  Interventions: Drug: ABT-354; Drug: Placebo
- Group 2, high dose (Experimental): ABT-354
  Interventions: Drug: ABT-354; Drug: Placebo

INTERVENTIONS:
Drug: ABT-354 — ABT-354 Low Dose
  Arms: Group 1, low dose
Drug: ABT-354 — ABT-354 High Dose
  Arms: Group 2, high dose
Drug: Placebo — Placebo

SUMMARY:
This study will investigate safety, tolerability and pharmacokinetics of ABT-354 in up to 20 male and female subjects, between 55 to 90 years of age with mild to moderate Alzheimer's disease on stable doses of acetylcholinesterase inhibitors.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, multiple-dose, multicenter study. Up to 20 male and female subjects with mild to moderate Alzheimer's disease (AD) who are taking stable doses of acetylcholinesterase inhibitors will be enrolled in this study. Within 28 days prior to study drug administration, subjects will be screened based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for probable AD, Mini-Mental State Examination (MMSE) and Modified Hachinski Ischemic Scale (MHIS) scores, medical history, physical examination, neurological examination, vital signs, ECG, laboratory tests and response to Columbia-Suicide Severity Rating Scale (C-SSRS).

The study will be performed in two groups of 10 subjects each. In each group of 10 subjects, 7 subjects will be randomly assigned to receive ABT-354 and 3 subjects to receive matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meets the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association criteria for probable Alzheimer's Disease
* Has a Mini-Mental State Examination total score of 16 to 26, inclusive, at Screening
* Has a Modified Hachinski Ischemia Scale score of ≤ 4 at Screening
* On a stable dose of - donepezil, galantamine or rivastigmine for at least 30 days prior to study drug administration
* Has had a computerized tomography or magnetic resonance imaging scan, interpreted by a radiologist or neurologist, within 36 months prior to randomization

Exclusion Criteria:

* Receipt of any depot drug by injection within 30 days prior to study drug administration
* Receipt of an investigational product within a time period equal to 10 half-lives, if known, or within 6 weeks prior to study drug administration
* History of any significant neurological disease other than Alzheimer's Disease
* History of significant sensitivity or allergy to multiple drugs based on medical records and/or the opinion of the investigator
* Significant current - suicidal ideation within 1 month prior to study drug administration as evidenced by answering "yes" to questions 4 or 5 on the suicidal ideation portion of the Columbia-Suicide Severity Rating Scale completed at Screening or any history of suicide attempts

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Vital signs | Up to Day 10
ECG (electrocardiogram) | Up to Day 10
Neurological exam | Up to Day 10
Laboratory tests | Up to Day 10
  Hematology, Chemistry, Urinalysis
Number of subject with adverse events | Up to Day 10
C-SSRS (Columbia-Suicide Severity Rating Scale) | Up to Day 10

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Up to Day 10
  Cmax, Cmin, Tmax, AUC, t-1/2, CL/F

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Marek, MD, Study Director — AbbVie
Locations (3):
- United States (3):
  - Site Reference ID/Investigator# 106999, Miami, Florida
  - Site Reference ID/Investigator# 106998, Orlando, Florida
  - Site Reference ID/Investigator# 107000, Overland Park, Kansas